CLINICAL TRIAL: NCT03568032
Title: The Clinical Study of Radiation-associated Carotid Artery Disease in Patients With Nasopharyngeal Carcinoma Treated by IMRT
Brief Title: Radiation-associated Carotid Artery Disease in Patients With Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiayun He, MD, Principal Investigator, Clinical Professor, Fudan University
Other Study IDs: NPC-CAROTID-01
Record Dates: First submitted 2018-03-29; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Nasopharyngeal Carcinoma; Carotid Artery Diseases
Keywords: intima media thickness
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the post-radiation group: patients diagnosed as non-metastatic nasopharyngeal carcinoma who received definitive IMRT more than 3 years ago
  Interventions: Diagnostic Test: Measurement of intima media thickness of carotid artery; Diagnostic Test: Detection and measurement of carotid plaques; Diagnostic Test: Carotid Color Flow Duplex Testing; Diagnostic Test: Montreal Cognitive Assessment; Other: Medical history of cardiovascular risk factors and cardiovascular diseases
- the pre-radiation group: untreated patients diagnosed as non-metastatic nasopharyngeal carcinoma
  Interventions: Diagnostic Test: Measurement of intima media thickness of carotid artery; Diagnostic Test: Detection and measurement of carotid plaques; Diagnostic Test: Carotid Color Flow Duplex Testing; Diagnostic Test: Montreal Cognitive Assessment; Other: Medical history of cardiovascular risk factors and cardiovascular diseases

INTERVENTIONS:
Diagnostic Test: Measurement of intima media thickness of carotid artery — IMT measurements were performed using ultrasound machine in the pre-radiation and the post-radiation group. IMT was assessed at the common carotid artery (CCA) and the internal carotid artery (ICA) of both the left and right side.
Diagnostic Test: Detection and measurement of carotid plaques — Detection and measurement of plaques within internal carotid artery and common carotid artery by ultrasound
Diagnostic Test: Carotid Color Flow Duplex Testing — Velocity measurement of carotid artery to determine carotid stenosis
Diagnostic Test: Montreal Cognitive Assessment — Cognitive assessment
Other: Medical history of cardiovascular risk factors and cardiovascular diseases — Cardiovascular risk factors include smoking, alcohol consumption, hypertension, diabetes mellitus, hypercholesterolemia, obesity. Cardiovascular diseases include ischemic stroke, ischemic coronary heart disease, TIA, etc.

SUMMARY:
Radiation-associated carotid vasculopathy is a common late sequelae in patients with head and neck cancer, which correlates with the incidence of stroke. Currently, little is known about the incidence of radiation-associated carotid vasculopahty in the context of intensity-modulated radiation therapy (IMRT).

The aim of this study is to determine whether IMRT will increase the incidence of carotid vasculopathy in patients with nasopharyngeal carcinoma (NPC).

ELIGIBILITY:
Inclusion Criteria:

* signed inform consent
* age more than 18 years old
* ECOG 0-2
* pathologic diagnosed, non-metastatic NPC
* either untreated or treated by definitive IMRT 3 years ago
* did not receive radiation to the head and neck region prior to the diagnosis of NPC
* if the patient received definitive IMRT 3 years ago because of NPC, he or she did not receive a second course of radiation due to local relapse
* no prior surgery of head and neck

Exclusion Criteria:

* prior history of cardiovascular disease before the diagnosis of NPC
* prior radiation to head and neck before the diagnosis of NPC
* prior surgery of head and neck
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is selected from new patients or post-radiation patients who come to the clinics of radiation oncology.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
intima media thickness of carotid artery | This is a cross-sectional study. So the time frame is within one week of a patient-visit to the clinics.
  the intima media thickness of common carotid artery, internal carotid artery of the left or right side

SECONDARY OUTCOMES:
the incidence of carotid stenosis | This is a cross-sectional study. So the time frame is within one week of a patient-visit to the clinics.
  Carotid stenosis is defined as the axial diameter of the carotid lumina decreases more than 50%.
the number of carotid plaques | This is a cross-sectional study. So the time frame is within one week of a patient-visit to the clinics.
  Carotid plaque is defined as a focal structure that encroaches into the arterial lumen of at least 0.5 mm or 50% of the surrounding IMT value or demonstrates a thickness >1.5 mm as measured from the media-adventitia interface to the intima- lumen interface.
total number of Montreal Cognitive Score (range: 0-30) | This is a cross-sectional study. So the time frame is within one week of a patient-visit to the clinics.
  the higher the number, the better the cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Xiayun He, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided